CLINICAL TRIAL: NCT03483662
Title: Dissemination and Implementation of the SPRINT Study Findings in Underserved Populations
Brief Title: Implementation of Multifaceted Patient-Centered Treatment Strategies for Intensive Blood Pressure Control (IMPACTS)
Acronym: IMPACTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jiang He, MD, PhD, Professor and Director, Tulane University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HL133790 (NIH); R01HL133790 (NIH)
Record Dates: First submitted 2018-03-24; First posted 2018-03-30 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2023-08

CONDITIONS: Hypertension; Blood Pressure
Keywords: hypertension; blood pressure; medication adherence; lifestyle modification; blood pressure control; implementation
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multicomponent Intervention (Experimental): Protocol-based treatment using the SPRINT stepped-care intensive BP management algorithm, dissemination of SPRINT study findings among provider-teams, patients, and administrators, team-based collaborative care, BP audit and feedback, home BP monitoring, and health coaching on antihypertensive medication adherence and lifestyle modification
  Interventions: Behavioral: Multicomponent Intervention
- Enhanced Usual Care (Active Comparator): Webinar education session for providers on the new ACC/AHA hypertensive clinical guideline and the SPRINT study findings
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Multicomponent Intervention — The core component of the intervention is protocol-based treatment using the SPRINT BP management algorithm. The following implementation strategies are adaptable components that will be modified to fit specific federally-qualified health center (FQHC) settings: dissemination of SPRINT study findings among provider-teams, patients, and administrators, team-based collaborative care, BP audit and feedback, home BP monitoring, and health coaching on antihypertensive medication adherence and lifestyle modification.
  Arms: Multicomponent Intervention
Behavioral: Enhanced Usual Care — The investigators will provide an up-to-date clinical guideline for hypertension management to providers. A webinar education session on the new American College of Cardiology (ACC)/American Heart Association (AHA) hypertension guideline and findings from the SPRINT trial will be conducted. Otherwise, the investigators will not conduct any active intervention and all control clinics will follow their routine clinic practice in the management of hypertensive patients
  Arms: Enhanced Usual Care

SUMMARY:
The IMPACTS study utilizes an effectiveness-implementation hybrid type 2 design to achieve two primary goals simultaneously: 1). to test the effectiveness of a multifaceted implementation strategy for intensive BP control among underserved hypertensive patients at high risk for CVD, and 2). to assess the implementation outcomes of the multifaceted implementation strategy in patients and providers.

DETAILED DESCRIPTION:
Recently, the Systolic Blood Pressure Intervention Trial (SPRINT) reported that more intensive blood pressure (BP) treatment (target systolic BP<120 mm Hg) reduced major cardiovascular disease (CVD) by about 25% and all-cause mortality by about 27% compared to standard BP treatment (target systolic BP<140 mm Hg) among hypertensive patients aged ≥50 years. SPRINT clearly answered the question - Will lowering BP more than the currently recommended goal further reduce the risk of CVD and mortality? The next important question is how to implement a more intensive BP treatment program in real-world clinical practice, especially in underserved patients. The IMPACTS trial is an effectiveness-implementation hybrid trial to simultaneously test the effectiveness of a multicomponent intervention program for more intensive BP treatment and the feasibility and fidelity of implementing the program in underserved patients with hypertension in Louisiana and Mississippi. The Consolidated Framework for Implementation Research has been used to guide the development of the multicomponent intervention, including dissemination of SPRINT study findings among patients, providers and policymakers; team-based collaborative care using a stepped-care protocol adapted from the SPRINT intensive-treatment algorithm, BP audit and feedback, and home BP monitoring; and health coaching on antihypertensive medication adherence and lifestyle modification. The investigators will collaborate with 36 federally qualified health center clinics that serve low-income populations in Louisiana and Mississippi to recruit 1,260 trial participants and conduct the IMPACTS trial. The primary clinical outcome is the difference in mean change of systolic BP from baseline to 18 months. The fidelity of the intervention, measured by intensification of treatment by providers and adherence to medications in patients, will be the primary implementation outcome. This study will generate urgently needed data on effective and adoptable intervention strategies aimed at eliminating health disparities and reducing the BP-related disease burden in underserved populations in the US.

ELIGIBILITY:
Eligibility Criteria for Clinics:

* Affiliated with participating FQHCs and not sharing providers or nurses/pharmacists with other clinics.
* Predominantly managing underserved populations with health disparities (ethnic minorities, low-income groups, and residents of rural areas and inner cities).
* Having electronic medical record systems.
* Serving >200 hypertension patients (ICD-10-CM I10-I15) during the previous year.
* Not participating in other hypertension control programs.

Inclusion Criteria for Study Participants:

* Men or women aged ≥40 years who receive primary care from the participating FQHC clinics.
* Systolic BP ≥140 mmHg at two screening visits for those not taking antihypertensive medication or systolic BP ≥ 130 mmHg at two screening visits for those taking antihypertensive medications.

Exclusion Criteria for Study Participants:

* Not able to understand English
* Pregnant women, women planning to become pregnant in the next 18 months, women of childbearing potential and not practicing birth control, and persons who cannot give informed consent.
* Plans to change to a primary healthcare provider outside of the FQHC clinic during the next 18 months.
* Diagnosis of end-stage renal disease, defined as dialysis or transplantation.
* Individuals unlikely to complete the study, such as those who plan to move out the study area during the next 18 months, temporary migrant workers, and homeless persons.
* Patients with immediate family members who are staff at their FQHC clinic.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1272 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Difference in mean change of systolic BP | Baseline to 18 months
  The primary outcome is the difference in mean change of systolic blood pressure from baseline to 18 months between intervention and control groups. Blood pressure will be measured 3 times each at two baseline, one 6-month, one 12-month, and two termination visits according to a standard protocol.
Difference in a fidelity summary score for key implementation strategy components during the 18-month intervention. | Baseline to 18 months
  A fidelity summary score includes adherence to antihypertensive medications, initiation or intensification of treatment, home BP monitoring, and health education over the intervention period. The fidelity summary score ranges from 0 (worst) to 4 (best)

SECONDARY OUTCOMES:
Proportion of patients with systolic blood pressure <120 mm Hg | Baseline to 18 months
  The differences in the proportion of patients with systolic blood pressure <120 mm Hg between the intervention and control groups at 18 months will be assessed.
Proportion of patients with systolic blood pressure <130 mm Hg | Baseline to 18 months
  The differences in the proportion of patients with systolic blood pressure <130 mm Hg between the intervention and control groups at 18 months will be assessed.
Proportion of patients with a >30 mm Hg reduction in systolic blood pressure | Baseline to 18 months
  The differences in the proportion of patients with a >30 mm Hg reduction in systolic blood pressure between the intervention and control groups at 18 months will be assessed.
Difference in mean change of diastolic blood pressure | Baseline to 18 months
  The difference in mean change of diastolic blood pressure from baseline to 18 months between intervention and control groups will be assessed.
Health-related quality of life (SF-12) | Baseline to 18 months
  Health-related quality of life will be assessed using the 12-Item Short Form Survey (SF-12). Physical component summary (PCS-12) and mental component summary (MCS-12) scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Intensification of treatment (fidelity) | Baseline to 18 months
  Survey data and electronic health record data will be used to assess whether providers add new antihypertensive medications or titrate existing medications. Intensification of antihypertension treatment is a binary outcome variable, with 1 representing the initiation of a new medication or an increase in the current medication dosage, and 0 representing no change in medication.
Medication adherence (fidelity) | Baseline to 18 months
  Patient medication adherence will be assessed by questionnaire. Binary variable: 1=high adherence and 0=low adherence
Self-reported home BP monitoring (fidelity) | Baseline to 18 months
  Patient home BP monitoring will be assessed by questionnaire. Binary variable: 1=yes and 0=no
Self-reported health education at previous clinic visits (fidelity) | Baseline to 18 months
  Patient health education at previous clinic visits will be assessed by questionnaire. Binary variable: 1=yes and 0=no.
Satisfaction with antihypertensive medications | Baseline to 18 months
  The satisfaction of patients with antihypertensive medications was assessed at baseline and follow-up visits using the question, 'How satisfied are you with antihypertensive medications you have received?' There are five possible answers: 'very satisfied,' 'satisfied,' 'neutral,' 'dissatisfied,' and 'very dissatisfied'.
Satisfaction with BP-related care | Baseline to 18 months
  The satisfaction of patients with BP-related care was assessed at baseline and follow-up visits using the question, 'How satisfied are you with the care you have received for your blood pressure?' There are five possible answers: 'very satisfied,' 'satisfied,' 'neutral,' 'dissatisfied,' and 'very dissatisfied'.
Acceptance to intensive BP target by providers in intervention clinics | Baseline to 18 months
  Survey among providers
Adherence to clinical appointments in the intervention group | Baseline to 18 months
  Study administrative data
Adherence to health coach session in the intervention group | Baseline to 18 months
  Study administrative data

CONTACTS AND LOCATIONS:
Overall Officials: Jiang He, MD, PhD, Principal Investigator — Tulane University; Marie A Krousel-Wood, MD, MPH, Principal Investigator — Tulane University
Locations (2):
- United States (2):
  - 26 FQHC Primary Care Clinics in Louisiana, New Orleans, Louisiana
  - 10 FQHC Primary Care Clinics in Mississippi, Biloxi, Mississippi

IPD SHARING:
Plan to Share IPD: Yes
The study data sharing plan will comply with all NIH policies for data sharing. Data sharing will be executed through the centralized NIH data repository. The study data will be prepared for transmission to the NHLBI data repository - the Biologic Specimen and Data Repository Information Coordinating Center. These data will be free of identifiers that allow identification of individual research participants either directly or through "deductive disclosure." At the completion of the project, the investigators will make all intervention materials and procedure manuals available to the public according to the approved plan for making data and materials available to the scientific community, lay public, and the NIH.
Supporting Information: Study Protocol
Time Frame: The data sets will be submitted to the study NHLBI study Program Official no later than 3 years after the end of the final patient follow-up or 2 years after the main paper of the trial has been published, whichever comes first.
Access Criteria: The investigators will offer, through our public access website, opportunities for outside investigators to collaborate with us using complete study data.

REFERENCES:
- [Derived] Mills KT, Peacock E, Chen J, Zimmerman A, He H, Cyprian A, Davis G, Fuqua SR, Gilliam DS, Greer A, Gray-Winfrey L, Williams S, Wiltz GM, Winfrey KL, Whelton PK, Krousel-Wood M, He J. Experiences and Beliefs of Low-Income Patients With Hypertension in Louisiana and Mississippi During the COVID-19 Pandemic. J Am Heart Assoc. 2021 Feb 2;10(3):e018510. doi: 10.1161/JAHA.120.018510. Epub 2020 Dec 3. PMID 33267723
- [Derived] Mills KT, Peacock E, Chen J, Zimmerman A, Brooks K, He H, Cyprian A, Davis G, Fuqua SR, Greer A, Gray-Winfrey L, Williams S, Wiltz GM, Winfrey KL, Whelton PK, Krousel-Wood M, He J. Implementation of Multifaceted Patient-Centered Treatment Strategies for Intensive Blood Pressure Control (IMPACTS): Rationale and design of a cluster-randomized trial. Am Heart J. 2020 Dec;230:13-24. doi: 10.1016/j.ahj.2020.08.009. Epub 2020 Aug 19. PMID 32827458